CLINICAL TRIAL: NCT05205291
Title: Molecular Imaging of LPS-induced Microglial Activation in Parkinson's Disease (PD). A TSPO PET-MR Imaging Study
Brief Title: Molecular Imaging of Inflammation in Parkinson's Disease Using LPS and TSPO-PET/MR
Status: Recruiting | Type: Observational
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 289952
Record Dates: First submitted 2021-11-09; First posted 2022-01-25 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Neurodegenerative Diseases; Parkinson Disease; REM Sleep Behavior Disorder (iRBD)
Keywords: Positron Emission Tomography; Inflammation; Neuroimaging; Biomarkers
MeSH Terms: conditions — Neurodegenerative Diseases; Parkinson Disease; REM Sleep Behavior Disorder; Inflammation | interventions — Lipopolysaccharides; (methyl-(11)C)N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The investigators will collect and retain venous blood samples for the analysis of inflammatory molecules (interleukines, chemokines, etc) to correlate with the imaging and clinical findings in patients with Parkinson's disease and healthy volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Parkinson's disease patients: 18 patients with Parkinson's disease who will undergo clinical assessment, and PET/MR imaging of TSPO using the tracer [11C]PBR28 before and four hours after administration of LPS (1 ng/Kg)
  Interventions: Drug: Lipopolysaccharide; Radiation: PET/MR with [11C]PBR28
- Healthy controls: 6 healthy controls who will undergo clinical assessment, and PET/MR imaging of TSPO using the tracer [11C]PBR28 before and four hours after administration of LPS (1 ng/Kg)
  Interventions: Drug: Lipopolysaccharide; Radiation: PET/MR with [11C]PBR28
- Patients with isolated REM sleep behavior disorder: Patients with a recent diagnosis of REM sleep behavior disorder

INTERVENTIONS:
Drug: Lipopolysaccharide — All participants will receive one dose of Lipopolysaccharide (1ng/Kg) after the first PET/MR scan with [11C]PBR28 and four hours before the second PET/MR scan with [11C]PBR28.
  Other Names: there is no other intervention
  Groups: Healthy controls; Parkinson's disease patients
Radiation: PET/MR with [11C]PBR28 — A PET/MR scan using the tracer [11C]PBR28 will be performed to all participants before and four hours after the administration of LPS
  Other Names: there is no other intervention
  Groups: Healthy controls; Parkinson's disease patients

SUMMARY:
It is not known what causes Parkinson's disease and what makes it worsen over time. Research conducted in the past few years has highlighted the possible role of inflammation on this process but its actual mechanisms are still obscure.

In this study, the investigators aim to gain understanding on how inflammation is increased in Parkinson's disease and what are its mechanisms, by performing two Positron Emission Tomography (PET) scans using the tracer [11C]PBR28, that takes pictures of the brain highlighting the areas of inflammation, before and after the administration of a compound called Lipopolysaccharide or LPS, that is known to cause a mild degree of inflammation. The investigators will couple this study with two venous blood draws to measure the levels of circulating molecules of inflammation.

DETAILED DESCRIPTION:
This is a cross-sectional study.

The study will be divided in two visits, of which, the visit 1 will take place in Exeter, and visit 2 will take place in London.

During visit 1, the participants will attend the NIHR Clinical Research Facility of Royal Devon & Exeter NHS Foundation Trust. The study doctor will explain all study procedures in a lay language and will answer all the participants' queries. After that, if they agree to participate, they will sign the informed consent. After this procedure, the study doctor will ask a few questions and assess whether the participant is suitable to be enrolled in the study. Then, the study doctor will undertake a clinical examination, and make some tests (questionnaires) to assess the presence of symptoms related to movement, thinking, memory, and behaviour. Finally, the study doctor will collect some blood and urine, for safety laboratory exams. Women of childbearing potential will also have a pregnancy test, for safety in view of the PET scans. After these procedures, the participants will be accompanied to the Mireille Gillings Neuroimaging Centre, that lies just opposite the Clinical Research Facility, and where they will perform the MRI scan. The MRI scan will collect pictures of the brain and will serve to gather information about the structure of the brain of the patients, and to exclude the concomitant presence of any lesion (incidental findings). The whole duration of the visit will be of around 3 hours, also counting the time for taking the consent and for the MRI scan.

During visit 2, the participants will attend the NIHR Imperial Clinical Research Facility and Invicro, in West London, over two consecutive days.

In the first day, the participants will attend the NIHR Imperial Clinical Research facility for a clinical visit to assess any change in medication or any side effect. Patients with Parkinson's disease will answer a few questionnaires on presence of symptoms related to PD. If more than 60 days have passed from the screening visit, participants will repeat the urine collection for safety analysis.

The participants (and one companion, if needed) will then be accompanied to the accommodation for the night, that is located just next to the MIHR Imperial Clinical Research Facility.

In the second day, the participants will attend Invicro for the PET visit. Invicro is a specialized centre for research on neuroimaging and is located opposite the accommodation facility. They will undergo a venous cannulation (for the injection of the tracer for the PET scans and for the injection of LPS) and an arterial cannulation (to collect some blood during the PET scans, that will serve to help with the analysis of the scans). the first PET scan will take place in the morning. After the PET scan, the participant will undergo the administration of LPS at the dose of 1 ng/Kg. Since LPS can cause side effects linked to neuroinflammation, the patient will have the blood pressure, heart rate, respiratory rate, and cardiac rhythm monitored for six hours, that is the mean duration of the effect of LPS. After four hours from the injection of LPS, the participants will undergo a second PET scan. The whole duration of the visit will be of around 8 hours. At the end of this visit, a sample of blood will be collected to repeat the safety laboratory tests. After this visit, the participants will be asked to attend the NIHR Imperial Clinical Research Facility for an overnight stay to monitor for any side effect, under medical supervision by a qualified doctor on call. After the overnight stay, if there won't be any side effect, the participant can be discharged and will have finished the study.

ELIGIBILITY:
Inclusion Criteria (all):

* 50-85 years of age, male or female
* Able to give informed consent
* Adequate visual and auditory acuity to complete the neuropsychological testing
* No presence or history of significant neurological or psychiatric disorders
* BDI ≥ 20, moderate depression
* No presence or history of inflammatory or autoimmune disorders
* Negative family history for neurodegenerative diseases
* Cognitively healthy (i.e., education-adjusted MoCA total score ≥ 26 points at screening)
* Female subjects must either be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or post-menopausal for at least 1 year (no menses for 12 months without an alternative medical cause) or if they are of childbearing potential, they must commit to use of a highly effective contraceptive measure for the duration of the study and a minimum of six months following the PET scan (including combined [estrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, or transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, or implantable], intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner or sexual abstinence).
* Male subjects and their partners of childbearing potential must commit to the use of a highly effective method of contraception during the study and for a minimum of three months following each PET scan (including, for female partners of childbearing potential, combined [estrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, or transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, or implantable], intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, male subjects with vasectomy or sexual abstinence).
* Male subjects must commit to not donate sperm during the study and for a minimum of three months after the last PET scan.
* Individuals must commit to refrain from drinking alcohol for 48 hours before each visit, refrain from drinking any caffeinated substance for 12 hours before the PET-MR visits, and to refrain from smoking or using any nicotine-containing products on the day of the PET-MR scans.
* Individuals must commit to not donating blood up to three months after the last PET scan.
* Individuals must commit to come to the screening and Day 1 visits in a fasting state (i.e., minimum of 8 hours since last meal/food intake).
* Individuals must commit to not to take any over-the-counter non-steroidal anti-inflammatory drugs or drink alcohol for 48h before screening visit.

Inclusion Criteria (Parkinson's disease patients):

* 50-85 years of age, male or female
* Able to give informed consent
* Adequate visual and auditory acuity to complete the neuropsychological testing
* No presence or history of other significant neurological or psychiatric disorders
* Diagnosis of PD according to the Movement Disorder Society Clinical Diagnostic Criteria (Postuma et al., Mov Disord 2015)
* Drug-naïve participants with PD must have a diagnosis of PD but must be therapy-free at the time of enrolment
* For participants with PD-MCI: diagnosis of MCI according the diagnostic criteria for MCI-PD (Level I; Litvan et al., Mov Disord 2012) and/or MoCA < 23
* For participants with PD taking dopaminergic therapy: must be in stable therapy (i.e. not have changed therapy in the last 60 days)
* Female subjects must either be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or post-menopausal for at least 1 year (no menses for 12 months without an alternative medical cause) or if they are of childbearing potential, they must commit to use of a highly effective contraceptive measure for the duration of the study and a minimum of six months following the PET scan (including combined [estrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, or transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, or implantable], intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner or sexual abstinence).
* Male subjects and their partners of childbearing potential must commit to the use of a highly effective method of contraception during the study and for a minimum of three months following each PET scan (including, for female partners of childbearing potential, combined [estrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, or transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, or implantable], intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, male subjects with vasectomy or sexual abstinence).
* Male subjects must commit to not donate sperm during the study and for a minimum of three months after the last PET scan.
* Individuals must commit to refrain from drinking alcohol for 48 hours before each visit, refrain from drinking any caffeinated substance for 12 hours before the PET-MR visits, and to refrain from smoking or using any nicotine-containing products on the day of the PET-MR scans.
* Individuals must commit to not donating blood up to three months after the last PET scan.
* Individuals must commit to come to the screening and Day 1 visits in a fasting state (i.e., minimum of 8 hours since last meal/food intake).
* Individuals must commit to not to take any over-the-counter non-steroidal anti-inflammatory drugs or drink alcohol for 48h before screening visit.

For participants with iRBD:

Inclusion criteria:

* 40-85 years of age, male or female
* Able to give informed consent
* Adequate visual and auditory acuity to complete the neuropsychological testing
* No presence or history of significant neurological or psychiatric disorders
* BDI-II ≥ 20, moderate depression
* No presence or history of inflammatory or autoimmune disorders
* Negative family history for neurodegenerative diseases
* Cognitively healthy (i.e., education-adjusted MoCA total score ≥ 26 points at screening)
* Female subjects must either be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or post-menopausal for at least 1 year (no menses for 12 months without an alternative medical cause) or if they are of childbearing potential, they must commit to use of a highly effective contraceptive measure for the duration of the study and a minimum of six months following the PET scan (including combined [estrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, or transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, or implantable], intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner or sexual abstinence).
* Male subjects and their partners of childbearing potential must commit to the use of a highly effective method of contraception during the study and for a minimum of three months following each PET scan (including, for female partners of childbearing potential, combined [estrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, or transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, or implantable], intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, male subjects with vasectomy or sexual abstinence).
* Male subjects must commit to not donate sperm during the study and for a minimum of three months after the last PET scan.
* Individuals must commit to refrain from drinking alcohol for 48 hours before each visit, refrain from drinking any caffeinated substance for 12 hours before the PET-MR visits, and to refrain from smoking or using any nicotine-containing products on the day of the PET-MR scans.
* Individuals must commit to not donating blood up to three months after the last PET scan.
* Individuals must commit to come to the screening and Day 1 visits in a fasting state (i.e., minimum of 8 hours since last meal/food intake).
* Individuals must commit to not to take any over-the-counter non-steroidal anti-inflammatory drugs or drink alcohol for 48h before screening visit.

Exclusion Criteria (all):

* Unwilling and/or unable to cooperate with study procedures
* Current or a recent (<12 months) history of drug or alcohol abuse/dependence
* BDI ≥ 20, moderate depression
* Presence of clinically significant (as deemed by the study physician) alterations on safety laboratory blood and urine testing
* Presence of comorbidities or concomitant medications incompatible with the assessment or imaging procedures as deemed by the study physician
* Recent (less than 30 days) use of antipsychotics and corticosteroids
* Recent (less than 2 days) use of NSAIDs.
* Use of any long-acting benzodiazepines (e.g., diazepam) or use of slow or medium acting benzodiazepines with doses ≥ 30 mg within 30 days prior to the first imaging scan.
* Presence of rs6971 genotype of low-affinity binders that hinders the measure of microglial activation with [11C]PBR28 PET
* Presence of neurological disorders and known intracranial co-morbidities such as stroke, haemorrhage, space-occupying lesions, signs of inflammation of the CNS
* Presence of serology compatible with HIV, syphilis, SARS-CoV2, or viral hepatitis
* History of autonomic dysfunction, previous vasovagal syncope or a positive tilt-test, and with bradycardia or use of medications causing bradycardia (e.g. beta-blockers)
* Pregnancy or breastfeeding
* Contraindication to MRI, such as presence of metal devises or implants, metal deposited in the body, or metal grains in the eyes
* History of cancer within the last 5 years, except for appropriately treated, non-melanoma skin carcinoma, non-metastatic prostate cancer, treated carcinoma in situ of the cervix or Stage I uterine cancer.
* Claustrophobia or history of back pain that makes prolonged laying on the PET or MRI scanner intolerable
* Contraindication to arterial cannulation, such as history of bleedings, haemorrhage, etc.
* Negative Allen's test (i.e. absence of collateral flow on hands on the test)
* Recent (less than 30 days) infection or vaccination (e.g. flu, SARS-CoV2 etc.)
* Concurrent participation to any clinical trial testing investigational drugs

Exclusion Criteria (Parkinson's disease patients):

* Unwilling and/or unable to cooperate with study procedures
* Current or recent history of drug or alcohol abuse/dependence
* BDI ≥ 20, moderate depression
* Presence of clinically significant (as deemed by the study physician) alterations on safety laboratory blood or urine testing
* Presence of comorbidities or concomitant medications incompatible with the assessment or imaging procedures as deemed by the study physician
* Recent (less than 30 days) use of antipsychotics and corticosteroids.
* Recent (less than 2 days) use of NSAIDs.
* Use of any long-acting benzodiazepines (e.g., diazepam) or use of slow or medium acting benzodiazepines with doses ≥ 30 mg within 30 days prior to the first imaging scan.
* Presence of rs6971 genotype of low-affinity binders that hinders the measure of microglial activation with [11C]PBR28 PET
* Presence of other neurological disorders and known intracranial co-morbidities such as stroke, haemorrhage, space-occupying lesions, signs of inflammation of the CNS
* History of autonomic dysfunction, previous vasovagal syncope or a positive tilt-test, and with bradycardia or use of medications causing bradycardia (e.g. beta-blockers)
* Presence of serology compatible with HIV, syphilis, SARS-CoV2, or viral hepatitis
* Pregnancy or breastfeeding
* Contraindication to MRI, such as presence of metal devises or implants, metal deposited in the body, or metal grains in the eyes
* History of cancer within the last 5 years, except for appropriately treated, non-melanoma skin carcinoma, non-metastatic prostate cancer, treated carcinoma in situ of the cervix or Stage I uterine cancer.
* Claustrophobia or history of back pain that makes prolonged laying on the PET or MRI scanner intolerable
* Contraindication to arterial cannulation, such as history of bleedings, haemorrhage, etc.
* Negative Allen's test (i.e. absence of collateral flow on hands on the test)
* Recent (less than 30 days) infection or vaccination (e.g. flu, SARS-CoV2 etc.)
* Concurrent participation to any clinical trial testing investigational drugs

Exclusion criteria (for participants with iRBD):

* Unwilling and/or unable to cooperate with study procedures
* Current or a recent (<12 months) history of drug or alcohol abuse/dependence
* BDI-II ≥ 20, moderate depression
* Presence of clinically significant (as deemed by the study physician) alterations on safety laboratory blood and urine testing
* Presence of comorbidities or concomitant medications incompatible with the assessment or imaging procedures as deemed by the study physician
* Recent (less than 30 days) use of antipsychotics and corticosteroids
* Recent (less than 2 days) use of NSAIDs.
* Use of any long-acting benzodiazepines (e.g., diazepam) or use of slow or medium acting benzodiazepines with doses ≥ 30 mg within 30 days prior to the first imaging scan.
* Use of any of the following drugs that might interfere with dopamine transporter SPECT imaging: Ephedrine, ketamine, isoflurane, cocaine, methylphenidate, amphetamine of any amphetamine derivatives, mazindol, modafinil, benztropine, fentanyl, derivatives, buproprion, phentermine neuroleptics, metoclopramide, alpha methyldopa, , reserpine, .
* Presence of rs6971 genotype of low-affinity binders that hinders the measure of microglial activation with [11C]PBR28 PET
* Presence of neurological disorders and known intracranial co-morbidities such as stroke, haemorrhage, space-occupying lesions, signs of inflammation of the CNS
* Presence of serology compatible with HIV, syphilis, or viral hepatitis
* History of autonomic dysfunction, previous vasovagal syncope or a positive tilt-test, and with bradycardia or use of medications causing bradycardia (e.g. beta-blockers)
* Pregnancy or breastfeeding
* Contraindication to MRI, such as presence of metal devises or implants, metal deposited in the body, or metal grains in the eyes
* History of cancer within the last 5 years, except for appropriately treated, non-melanoma skin carcinoma, non-metastatic prostate cancer, treated carcinoma in situ of the cervix or Stage I uterine cancer.
* Claustrophobia or history of back pain that makes prolonged laying on the PET or MRI scanner intolerable
* Contraindication to arterial cannulation, such as history of bleedings, haemorrhage, etc.
* Negative Allen's test (i.e. absence of collateral flow on hands on the test)
* Recent (less than 30 days) infection or vaccination (e.g. flu, SARS-CoV2 etc.)
* Evidence of presynaptic dopaminergic denervation on [123I]FP-CIT SPECT
* Concurrent participation to any clinical trial testing investigational drugs

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease: 18 in total, divided in early drug-naive Parkinson's disease (6); Parkinson's disease in pharmacological therapy(6); Advanced Parkinson's disease (6).
  Patients with REM sleep behavior disorder: 6 in total;
  Healthy volunteers (6).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in inflammation in the brain following administration of LPS | 36 months
  To evaluate whether the activation of microglia following administration of LPS, as measured with PET/MR and the tracer [11C]PBR28, is changed in patients with Parkinson's disease compared with healthy volunteers

SECONDARY OUTCOMES:
Correlation of LPS-induced increase of inflammation and cerebral perfusion | 36 months
  To evaluate whether the administration of LPS increases the cerebral perfusion, as measured with Arterial Spin Labelling (ASL) in patients with Parkinson's disease compared with healthy volunteers
Correlation of LPS-induced increase of inflammation and resting state functional MRI (rs fMRI) | 36 months
  To evaluate whether the administration of LPS changes resting state functional Magnetic Resonance Imaging (rs-fMRI) parameters, which measure the strength of functional connectivity in the brain, in patients with Parkinson's disease compared with healthy volunteers
Safety of LPS administration in Parkinson's disease patients | 36 months
  To evaluate whether the administration of LPS is safe to use as a paradigm of in vivo study of inflammation in patient with Parkinson's disease, as measured by the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) and by overnight monitoring of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Marios Politis, MD MSc PhD, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No